CLINICAL TRIAL: NCT01545297
Title: Comparison of Dexmedetomidine and Propofol-Remifentanil Conscious Sedation for Awake Craniotomy for Tumor Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Dexmedetomidine and Propofol-Remifentanil Conscious Sedation for Awake Craniotomy for Tumor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Goettel (Other)
Responsible Party: Sponsor-Investigator, Nicolai Goettel, MD, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0607-A
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Brain Tumor
Keywords: dexmedetomidine; conscious sedation; awake craniotomy; brain mapping
MeSH Terms: conditions — Brain Neoplasms | interventions — Dexmedetomidine; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol-Remifentanil (Active Comparator): Group I. (propofol/remifentanil): Infusions begin at remifentanil (0.01-0.1 mcg/kg/min) and propofol (25-250 mcg/kg/min) for 15 min, and then titrated to effect.
  Interventions: Drug: Propofol; Drug: Remifentanil
- Dexmedetomidine (Experimental): Group II. (dexmedetomidine): The infusion begins at 0.3-0.4 mcg/kg/hr for 15 min, and then titrated down to 0.1-0.2 mcg/kg/hr.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The infusion begins at dexmedetomidine 0.3-0.4 mcg/kg/hr for 15 min, and then titrated down to 0.1-0.2 mcg/kg/hr.
  Other Names: Precedex (TM)
  Arms: Dexmedetomidine
Drug: Propofol — The infusion begins at propofol 25-250 mcg/kg/min for 15 min, and then titrated to effect.
  Other Names: Diprivan (TM)
  Arms: Propofol-Remifentanil
Drug: Remifentanil — The infusion begins at remifentanil 0.01-0.1 mcg/kg/min for 15 min, and then titrated to effect.
  Other Names: Ultiva (TM)
  Arms: Propofol-Remifentanil

SUMMARY:
Awake craniotomy for resection of brain tumor located in close proximity to areas of eloquent brain function, such as speech, motor and sensory, is an accepted procedure used to minimize neurological injury during resection. During awake craniotomy, anesthesia is usually provided using a combination of local anesthesia (regional scalp block and/or local infiltration) and intravenous (IV) agents to provide sedation, anxiolysis and analgesia. Propofol sedation, commonly in combination with a shorter acting opioid such as fentanyl, or remifentanil, is an effective and popular technique during awake craniotomy, achieving a high degree of patient satisfaction and acceptance. Most of the anesthetic agents are associated with some respiratory depression.

The anesthetic agent called dexmedetomidine is a potent, highly selective α2-adrenoceptor agonist. The effects of dexmedetomidine are anxiolysis, analgesia, sedation and sympatholysis, and it is not associated with respiratory depressive effect. Bekker et al. first reported the successful use of dexmedetomidine in awake craniotomy in 2001.

The purpose of this blinded, prospective, randomized study is to compare the efficacy of dexmedetomidine versus propofol-remifentanil based sedation in patients undergoing awake craniotomy for resection of tumors. The study hypothesis is that the efficacy of performing intra-operative brain mapping is identical between dexmedetomidine and the propofol-remifentanil based sedation. The primary end-points are to assess the ability to perform intraoperative mapping during awake craniotomy. Secondary end-points will assess the incidence of complications (respiratory depression, failure to provide adequate analgesia), as well as patient and surgeon satisfaction to the corresponding anesthetic technique.

DETAILED DESCRIPTION:
Awake craniotomy for resection of brain tumor located in close proximity to areas of eloquent brain function, such as speech, motor and sensory, is an accepted procedure used to minimize neurological injury during resection. The level of sedation and analgesia during the different stages of surgery varies, but importantly, the patient needs to be awake and alert during brain mapping. During awake craniotomy, anesthesia is usually provided using a combination of local anesthesia (regional scalp block and/or local infiltration) and intravenous (IV) agents to provide sedation, anxiolysis and analgesia. There is considerable variation in the anesthetic management of the awake craniotomy in different institutions. Propofol sedation, commonly in combination with a shorter acting opioid such as fentanyl, or remifentanil, is an effective and popular technique during awake craniotomy, achieving a high degree of patient satisfaction and acceptance. However, the awake craniotomy remains one of the most challenging techniques of anesthesia care in terms of balancing an adequate depth of sedation and analgesia to combat the rapid changes of surgical stimulation yet having an alert patient for brain mapping. Furthermore, most of the anesthetic agents are associated with some respiratory depression.

A newer anesthetic agent called dexmedetomidine (Precedex (TM), Hospira Healthcare Corporation, Saint Laurent, Québec, Canada) is a potent, highly selective α2-adrenoceptor agonist with an α2:α1 selectivity ratio of 1600:1. It has been available in the Canada since 2009 as a short-term sedative agent, and is available in the UHN. The use of dexmedetomidine has been in mechanically ventilated patients in ICU and for intra-operative sedation. The well-documented beneficial effects of dexmedetomidine are anxiolysis, analgesia, sedation and sympatholysis, and it is not associated with respiratory depressive effect.

Dexmedetomidine has been successfully used to provide sedation in dental procedures, awake fibreoptic intubation, bariatric surgery and morbidly obese patients, as well as obstructive sleep apnea patients. The pharmacokinetic properties of dexmedetomidine is very predictable and titratable, with a rapid distribution half-life (t1/2α) being approximately 5-6min and an elimination half-life (t1/2β) of approximately 2h. Bekker et al. first reported the successful use of dexmedetomidine in awake craniotomy in 2001. Subsequent case series published by Souter et al. demonstrated that dexmedetomidine can be used either as a sole agent or in combination with other agents such as fentanyl during seizure foci resection with accurate intraoperative brain mapping.

The hypnotic effect of dexmedetomidine is mediated by the hyperpolarization of noradrenergic neurons in the locus ceruleus, which proposed that dexmedetomidine converges on a natural sleep pathway to exert its sedative effect. Venn and co-workers, as part of a large European multicentre trial investigating dexmedetomidine for postoperative sedation in the ICU, reported that: "Patients are calmly and easily roused from sleep to allow excellent communication and cooperation while intubated and ventilated, and then similarly quickly return to sleep". This unique sedation state is very useful for awake craniotomy, which requires deep level of sedation during painful operative procedures, as well as easily rousable state during mapping of eloquent function.

The purpose of this blinded, prospective, randomized study is to compare the efficacy of dexmedetomidine versus propofol-remifentanil based sedation in patients undergoing awake craniotomy for resection of tumors. The study hypothesis is that the efficacy of performing intra-operative brain mapping is identical between dexmedetomidine and the propofol-remifentanil based sedation. The primary end-points are to assess the ability to perform intraoperative mapping during awake craniotomy. Secondary end-points will assess the incidence of complications (respiratory depression, failure to provide adequate analgesia), as well as patient and surgeon satisfaction to the corresponding anesthetic technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients more than 18 years of age.
* ASA score I, II and III.
* Patients scheduled to undergo awake craniotomy for elective tumor resection.

Exclusion Criteria:

* Patients with allergies to the drugs being used.
* Patients who are pregnant.
* Patients with alcohol or substance abuse.
* Patients who are not able to understand the instructions for an awake craniotomy and questions regarding intra-operative pain, and post-operative satisfaction.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Ability to perform intra-operative mapping during awake craniotomy | immediately, intra-operative

SECONDARY OUTCOMES:
Incidence of complications (respiratory depression, failure to provide adequate analgesia) | intra-operatively, 2h post-operatively, 24h post-operatively
Patient and surgeon satisfaction to the corresponding anesthetic technique | intra-opeartively, 2h post-operatively, 24h post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Manninen, MD, FRCPC, Principal Investigator — Head of Neuroanesthesia, Associate Professor, University Health Network, Department of Anesthesia, University of Toronto, Canada; Nicolai Goettel, MD, Study Director — University Health Network, Department of Anesthesia, University of Toronto, Canada
Locations (1):
- UHN Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Serletis D, Bernstein M. Prospective study of awake craniotomy used routinely and nonselectively for supratentorial tumors. J Neurosurg. 2007 Jul;107(1):1-6. doi: 10.3171/JNS-07/07/0001. PMID 17639865
- [Background] Blanshard HJ, Chung F, Manninen PH, Taylor MD, Bernstein M. Awake craniotomy for removal of intracranial tumor: considerations for early discharge. Anesth Analg. 2001 Jan;92(1):89-94. doi: 10.1097/00000539-200101000-00018. PMID 11133607
- [Background] Johnson KB, Egan TD. Remifentanil and propofol combination for awake craniotomy: case report with pharmacokinetic simulations. J Neurosurg Anesthesiol. 1998 Jan;10(1):25-9. doi: 10.1097/00008506-199801000-00006. PMID 9438615
- [Background] Berkenstadt H, Perel A, Hadani M, Unofrievich I, Ram Z. Monitored anesthesia care using remifentanil and propofol for awake craniotomy. J Neurosurg Anesthesiol. 2001 Jul;13(3):246-9. doi: 10.1097/00008506-200107000-00013. PMID 11426102
- [Background] Sarang A, Dinsmore J. Anaesthesia for awake craniotomy--evolution of a technique that facilitates awake neurological testing. Br J Anaesth. 2003 Feb;90(2):161-5. doi: 10.1093/bja/aeg037. PMID 12538371
- [Background] Silbergeld DL, Mueller WM, Colley PS, Ojemann GA, Lettich E. Use of propofol (Diprivan) for awake craniotomies: technical note. Surg Neurol. 1992 Oct;38(4):271-2. doi: 10.1016/0090-3019(92)90038-o. PMID 1440214
- [Background] Coles JP, Leary TS, Monteiro JN, Brazier P, Summors A, Doyle P, Matta BF, Gupta AK. Propofol anesthesia for craniotomy: a double-blind comparison of remifentanil, alfentanil, and fentanyl. J Neurosurg Anesthesiol. 2000 Jan;12(1):15-20. doi: 10.1097/00008506-200001000-00004. PMID 10636615
- [Background] From RP, Warner DS, Todd MM, Sokoll MD. Anesthesia for craniotomy: a double-blind comparison of alfentanil, fentanyl, and sufentanil. Anesthesiology. 1990 Nov;73(5):896-904. PMID 1978615
- [Background] Manninen PH, Balki M, Lukitto K, Bernstein M. Patient satisfaction with awake craniotomy for tumor surgery: a comparison of remifentanil and fentanyl in conjunction with propofol. Anesth Analg. 2006 Jan;102(1):237-42. doi: 10.1213/01.ANE.0000181287.86811.5C. PMID 16368836
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Kamibayashi T, Maze M. Clinical uses of alpha2 -adrenergic agonists. Anesthesiology. 2000 Nov;93(5):1345-9. doi: 10.1097/00000542-200011000-00030. No abstract available. PMID 11046225
- [Background] Cheung CW, Ying CL, Chiu WK, Wong GT, Ng KF, Irwin MG. A comparison of dexmedetomidine and midazolam for sedation in third molar surgery. Anaesthesia. 2007 Nov;62(11):1132-8. doi: 10.1111/j.1365-2044.2007.05230.x. PMID 17924894
- [Background] Bamgbade OA, Alfa JA. Dexmedetomidine anaesthesia for patients with obstructive sleep apnoea undergoing bariatric surgery. Eur J Anaesthesiol. 2009 Feb;26(2):176-7. doi: 10.1097/EJA.0b013e32831a47cb. No abstract available. PMID 19142095
- [Background] Chawla S, Robinson S, Norton A, Esterman A, Taneerananon T. Peri-operative use of dexmedetomidine in airway reconstruction surgery for obstructive sleep apnoea. J Laryngol Otol. 2010 Jan;124(1):67-72. doi: 10.1017/S002221510999123X. Epub 2009 Oct 26. PMID 19852868
- [Background] Ramsay MA, Saha D, Hebeler RF. Tracheal resection in the morbidly obese patient: the role of dexmedetomidine. J Clin Anesth. 2006 Sep;18(6):452-4. doi: 10.1016/j.jclinane.2006.02.004. PMID 16980164
- [Background] Coursin DB, Coursin DB, Maccioli GA. Dexmedetomidine. Curr Opin Crit Care. 2001 Aug;7(4):221-6. doi: 10.1097/00075198-200108000-00002. PMID 11571417
- [Background] Bekker AY, Kaufman B, Samir H, Doyle W. The use of dexmedetomidine infusion for awake craniotomy. Anesth Analg. 2001 May;92(5):1251-3. doi: 10.1097/00000539-200105000-00031. No abstract available. PMID 11323355
- [Background] Souter MJ, Rozet I, Ojemann JG, Souter KJ, Holmes MD, Lee L, Lam AM. Dexmedetomidine sedation during awake craniotomy for seizure resection: effects on electrocorticography. J Neurosurg Anesthesiol. 2007 Jan;19(1):38-44. doi: 10.1097/01.ana.0000211027.26550.24. PMID 17198099
- [Background] Oda Y, Toriyama S, Tanaka K, Matsuura T, Hamaoka N, Morino M, Asada A. The effect of dexmedetomidine on electrocorticography in patients with temporal lobe epilepsy under sevoflurane anesthesia. Anesth Analg. 2007 Nov;105(5):1272-7, table of contents. doi: 10.1213/01.ane.0000281075.77316.98. PMID 17959954
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Venn RM, Bradshaw CJ, Spencer R, Brealey D, Caudwell E, Naughton C, Vedio A, Singer M, Feneck R, Treacher D, Willatts SM, Grounds RM. Preliminary UK experience of dexmedetomidine, a novel agent for postoperative sedation in the intensive care unit. Anaesthesia. 1999 Dec;54(12):1136-42. doi: 10.1046/j.1365-2044.1999.01114.x. PMID 10594409
- [Background] Conte V, Magni L, Songa V, Tomaselli P, Ghisoni L, Magnoni S, Bello L, Stocchetti N. Analysis of propofol/remifentanil infusion protocol for tumor surgery with intraoperative brain mapping. J Neurosurg Anesthesiol. 2010 Apr;22(2):119-27. doi: 10.1097/ANA.0b013e3181c959f4. PMID 20118799
- [Background] Mack PF, Perrine K, Kobylarz E, Schwartz TH, Lien CA. Dexmedetomidine and neurocognitive testing in awake craniotomy. J Neurosurg Anesthesiol. 2004 Jan;16(1):20-5. doi: 10.1097/00008506-200401000-00005. PMID 14676565
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- [Derived] Goettel N, Bharadwaj S, Venkatraghavan L, Mehta J, Bernstein M, Manninen PH. Dexmedetomidine vs propofol-remifentanil conscious sedation for awake craniotomy: a prospective randomized controlled trial. Br J Anaesth. 2016 Jun;116(6):811-21. doi: 10.1093/bja/aew024. Epub 2016 Apr 20. PMID 27099154